CLINICAL TRIAL: NCT04766424
Title: Effects of a Behavioral Sleep Extension Intervention on Cardiometabolic Risk Factors Among Patients With Elevated BP/Hypertension
Brief Title: Sleep Technology Intervention to Target Cardiometabolic Health
Acronym: STITCH
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: University of Illinois at Chicago (Other); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Kelly Glazer Baron, Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10055552; 1R01NR018891-01A1 (NIH)
Record Dates: First submitted 2021-02-13; First posted 2021-02-23 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Elevated Blood Pressure; Habitual Sleep Duration of Less Than or Equal to 7 Hours
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigators and outcomes assessors will not have access to the randomization table. Outcomes assessors will not be involved in the group assignments. Participants will be instructed to not tell outcomes assessors which group they are assigned to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral sleep extension group (Experimental): Participants in the sleep extension group will receive a fitbit, weekly coaching calls and educational materials for 8 weeks. In months 3-6, they will receive educational materials and an email from the coach each month.
  Interventions: Behavioral: Sleep extension intervention
- Health education (Other): Participants in the health education group will receive 8 weekly health education emails and telephone calls to confirm their receipt and clarify any concepts from the materials. In months 3-6, they will receive monthly health education materials.
  Interventions: Behavioral: Health education

INTERVENTIONS:
Behavioral: Sleep extension intervention — Participants will receive a fitbit and 8 weekly sleep-related educational materials via email and telephone coaching to review their sleep tracker data, set goals, trouble shoot any problems, and increase motivation.
  Arms: Behavioral sleep extension group
Behavioral: Health education — Participants will receive 8 weekly health education newsletters delivered via email.
  Arms: Health education

SUMMARY:
The goal of this study is to test the efficacy of a behavioral sleep extension intervention on sleep duration, cardio-metabolic disease risk factors, and health behaviors among adults with elevated blood pressure/hypertension and short sleep duration.

DETAILED DESCRIPTION:
Half of U.S. adults have at least one cardio-metabolic disease (CMD), including hypertension (HTN), heart disease, stroke, or diabetes. Even with advances in screening, education, and medication management, controlling these chronic diseases remains challenging. Despite the well-established negative effects of short sleep duration, surprisingly few studies have tested the benefits of sleep extension and even fewer studies evaluate the science of sleep extension interventions. Therefore, the goal of this study is to test the efficacy of a behavioral sleep extension intervention on sleep duration, CMD risk factors, and health behaviors among adults with elevated BP/HTN and short sleep duration.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* 24h ABP readings indicating elevated blood pressure (BP) or hypertension (24h average systolic (SBP) of 115-145 mmHg or diastolic (DBP) of 75-90 mmHg). Patients taking antihypertensive medications will be permitted if stable dose for >8 weeks
* Time in bed <8 hours and habitual sleep duration <7 hours via actigraphy;
* Smartphone user
* Able to read/write in English.

Exclusion Criteria:

* High risk or presence of moderate to severe comorbid sleep disorders (i.e., obstructive sleep apnea AHI 15 or greater, restless legs syndrome, or insomnia) as assessed by the questionnaires and overnight obstructive sleep apnea at the baseline/screening
* Resistant hypertension, defined as >4 antihypertensive medications or taking medications and standardized in lab BP >130 mmHg SBP or 80 mmHg DBP at screening History of cognitive or neurological disorders (e.g. dementia, Parkinson's, Multiple Sclerosis)
* BMI>50 kg/m2 or arm circumference greater than extra large cuff
* Presence of major psychiatric disorders (e.g. schizophrenia, bipolar disorder)
* alcohol abuse on the Audit-C (score >4 for men, >3 for women)
* drug use on the NIDA-Modified ASSIST (score >3),90
* moderate to severe depressive symptoms (PHQ-8 >10)
* Unstable or serious medical illness that would interfere with participation (cancer, renal disease on dialysis)
* Overnight work more than 1x per month
* Use of hypnotic or stimulant medications
* Situations that would significantly impact the ability to extend sleep, including overnight caregiving responsibility for children under the age 1, elderly or disabled adults >1x per week
* Inability to read or write in English
* Pregnancy/desire to become pregnant during the study period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2024-06-14 (Actual); Study Completion 2025-06-14 (Estimated)

PRIMARY OUTCOMES:
Sleep duration | 8 weeks
  Sleep duration will be measured using wrist actigraphy for 7 days

SECONDARY OUTCOMES:
24 hour ambulatory blood pressure | 8 weeks
  Ambulatory blood pressure glycemic control, lipids).
24 hour ambulatory blood pressure | 12 months
  Ambulatory blood pressure glycemic control, lipids).
Sleep duration | 12 months
  Sleep duration will be measured using wrist actigraphy for 7 days

OTHER OUTCOMES:
Diet | 8 weeks
  24 hour diet recall
Diet | 12 months
  24 hour diet recall
Physical activity | 8 weeks
  Accelerometer measured activity over 7 days
Physical activity | 12 months
  Accelerometer measured activity over 7 days
HbA1c | 12 months
  Cardiometabolic marker
C-reactive protein (CRP) | 8 weeks
  Cardiometabolic marker
C-reactive protein (CRP) | 12 months
  Cardiometabolic marker
IL-6 | 8 weeks
  Cardiometabolic marker
IL-6 | 12 months
  Cardiometabolic marker

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available upon request to the investigators at the end of the study.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within 1 year upon completion fo the study
Access Criteria: Written request to the PI

REFERENCES:
- [Derived] Baron KG, Duffecy J, Simonsen S, Bress A, Conroy MB, Greene T, Allen C, Vallejo S. Sleep Technology Intervention to Target Cardiometabolic Health (STITCH): a randomized controlled study of a behavioral sleep extension intervention compared to an education control to improve sleep duration, blood pressure, and cardiometabolic health among adults with elevated blood pressure/hypertension. Trials. 2023 Oct 10;24(1):658. doi: 10.1186/s13063-023-07658-6. PMID 37817267